CLINICAL TRIAL: NCT06783478
Title: Phase II Multicenter, Double-Blind, Prospective, Randomized Clinical Trial of NK Cell Infusion for Remission Consolidation in Patients With Acute Myeloid Leukemia
Brief Title: NK Cell Infusion for Remission Consolidation in AML: A Phase II Trial
Acronym: NKLMA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0533; D9A9CC97-F464-4C99-AC57-1E0E93 (Other Grant/Funding Number: FINEP)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukaemia (AML)
Keywords: Adoptive Immunotherapy; Natural Killer Cells; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Six infusions of 1 x 10⁷/kg of haploidentical NK cells, in vitro expanded and activated.
  Interventions: Biological: NK cell infusion
- Placebo (Placebo Comparator): Six infusions of placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NK cell infusion — Six infusions of 1 x 10⁷/kg of haploidentical NK cells, in vitro expanded and activated.
  Arms: Treatment
Other: Placebo — Six infusions of placebo
  Arms: Placebo

SUMMARY:
Acute Myeloid Leukemia (AML) is a complex and rapidly progressive disease with high mortality. Although significant progress has been made in recent years with the development of new drugs, resulting in better therapeutic tolerability and increased survival, disease relapse occurs in most cases. Adoptive immunotherapy has been increasingly emerging as an innovative alternative for cancer treatment. Among the immune cells tested, natural killer (NK) cells appear to exert significant antileukemic activity, particularly against AML, as demonstrated by numerous phase I/II studies published in the literature, including studies from our group.

This study aims to test whether haploidentical NK cells from healthy individuals, expanded and activated in vitro, administered when the disease is nearly eradicated by chemotherapy, can eliminate residual disease, delaying or eliminating the possibility of relapse. It is a randomized, superiority, double-blind, placebo-controlled clinical trial conducted at two treatment centers in Brazil. Adult patients aged 18 to 75 years with AML, from any risk group, in complete remission after completing standard treatment, will be included. Those with a bone marrow donor and eligible for this treatment will be allowed to undergo hematopoietic stem cell transplantation (HSCT). The study's objective is to determine whether the infusion of haploidentical NK cells immediately after high-dose chemotherapy results in increased event-free survival (EFS), overall survival (OS), and lower minimal residual disease (MRD) during follow-up or immediately before HSCT compared to patients undergoing the same treatment without NK cell infusion. A total of 98 participants in complete remission (CR) will be randomized to receive 6 infusions of 1 x 10⁷ NK cells/kg or 6 placebo infusions.

All participants will be evaluated for immune recovery at the cellular and molecular levels, and their immune profiles will be compared to analyze cellular response mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 59 years, and 60 to 75 years if their score is < 0.4 on the 10-minute Comprehensive Geriatric Assessment (CGA-10);
* Recently diagnosed acute myeloid leukemia, excluding acute promyelocytic leukemia confirmed by the molecular finding of PML-RARA or the presence of t(15:17) in genetic evaluation;
* In first complete hematologic remission after remission induction;
* Eligible, in the opinion of the principal investigator, to undergo consolidation chemotherapy with HDAra-C;
* No history of NYHA > III heart failure, acute myocardial infarction, or unstable angina in the past 6 months;
* Negative beta-HCG test for women of childbearing potential and agreement to use contraceptive methods throughout the treatment, from the time of informed consent signature until one month after the last dose of treatment;
* Non-reactive HIV serology;
* No prior investigational therapy in the 4 weeks before study enrollment;
* Availability of a haploidentical peripheral blood donor;
* Signed informed consent form.

Exclusion Criteria:

* Patients under 18 years of age; or aged 60 to 75 years with a score > 0.4 on the CGA-10 scale; or over 76 years of age, regardless of the score on the CGA-10 scale.
* Diagnosis of acute promyelocytic leukemia confirmed by the molecular finding of PML-RARA or the presence of t(15:17) in genetic evaluation.
* Failure to achieve first complete hematologic remission after remission induction.
* Ineligible, in the investigator's opinion, to undergo consolidation chemotherapy with HDAra-C.
* History of NYHA > III heart failure, acute myocardial infarction, or unstable angina in the past 6 months.
* Positive beta-HCG test for women of childbearing potential or non-compliance with using contraceptive methods throughout the treatment, from the time of informed consent signature until one month after the last dose of treatment.
* Reactive HIV serology.
* Prior investigational therapy in the four weeks preceding study enrollment.
* Lack of availability of a haploidentical peripheral blood donor.
* Failure to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 24 months

SECONDARY OUTCOMES:
Overall response rate (ORR) | 24 months
Pre-transplant minimal residual disease (MRD) measurement | The minimal residual disease (MRD) will be measured 4 weeks before the transplant for patients who will undergo hematopoietic stem cell transplantation (HSCT).
Immune Recovery | 24 months
Chimerism | 24 months
Depression Scale | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided